CLINICAL TRIAL: NCT05650918
Title: Dendritic Cells Loaded With Allogeneic Tumor Lysate (MesoPher) in Combination With a CD40 Agonist (Mitazalimab) in Metastatic Pancreatic Disease
Brief Title: MesoPher/Mitazalimab-combination Therapy in Metastatic Pancreatic Disease (REACtiVe-2 Trial)
Acronym: REACtiVe-2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joachim Aerts, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Joachim Aerts, MD PhD, Prof. dr., Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: NL76592.000.21
Record Dates: First submitted 2022-08-08; First posted 2022-12-14 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: Immunotherapy; CD40 agonist; Dendritic cell therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — mitazalimab

STUDY DESIGN:
Intervention Model Description: open-label, dose-finding, single-center phase I study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MesoPher and mitazalimab combination therapy (Experimental): MesoPher. 25 million lysate loaded DCs administered in the form of 3 biweekly and 2 additional vaccinations (3 and 6 months after the third vaccination). 1/3 intradermal injection in the forearm and 2/3 via the intravenous route.
  mitazalimab, 75µg/kg-150µg/kg-300µg/kg-600µg/kg or 1200µg/kg via intravenous route in the form of 3 biweekly and 2 additional infusions (3 and 6 months after the third vaccination).
  Interventions: Biological: MesoPher; Biological: Mitazalimab

INTERVENTIONS:
Biological: MesoPher — autologous monocyte-derived dendritic cells loaded with PheraLys (tumor cell lysate)
Biological: Mitazalimab — agonistic human monoclonal (IgG1) antibody targeting CD40

SUMMARY:
Pancreatic cancer is expected to be the second leading cause of cancer-related death in 2020. Pancreatic cancer is known as an immunological cold tumor. It is thought that the characteristic desmoplastic stroma of established pancreatic adenocarcinomas acts as a physical as well as an immunosuppressive barrier leading to exclusion of T cells. The use of CD40 agonists (such as mitazalimab, also known as JNJ-64457107 and ADC-1013) may convert pancreatic adenocarcinomas into immunological hot tumors by T-cell-dependent and T-cell-independent mechanisms. Targeting the desmoplastic stroma, thereby making the tumor more permeable for T-cell infiltration, is seen as one of the assisting mechanisms. Furthermore, the immunological coldness of pancreatic cancers infers that tumor-reactive T-cell responses are absent or weak at best. Dendritic cell therapy introduces tumor-specific T cells and in combination with a CD40 agonist, may lead to synergistic anti-tumor responses which could be beneficial for pancreatic cancer patients.

DETAILED DESCRIPTION:
Rationale: Pancreatic cancer is expected to be the second leading cause of cancer-related death in 2020. Pancreatic cancer is known as an immunological cold tumor. It is thought that the characteristic desmoplastic stroma of established pancreatic adenocarcinomas acts as a physical as well as an immunosuppressive barrier leading to exclusion of T cells. The use of CD40 agonists (such as mitazalimab, also known as JNJ-64457107 and ADC-1013) may convert pancreatic adenocarcinomas into immunological hot tumors by T-cell-dependent and T-cell-independent mechanisms. Targeting the desmoplastic stroma, thereby making the tumor more permeable for T-cell infiltration, is seen as one of the assisting mechanisms. Furthermore, the immunological coldness of pancreatic cancers infers that tumor-reactive T-cell responses are absent or weak at best. Dendritic cell therapy introduces tumor-specific T cells and in combination with a CD40 agonist, may lead to synergistic anti-tumor responses which could be beneficial for pancreatic cancer patients.

Objective: To investigate safety and tolerability as well as the induced immune response upon MesoPher/mitazalimab combination therapy in metastasized pancreatic cancer after standard-of-care (SOC) treatment with (modified) FOLFIRINOX.

Study design: Open-label, single-center, phase I dose finding study using a modified toxicity probability interval (mTPI) design.

Study population: Adults with metastatic pancreatic cancer after SOC treatment with (modified) FOLFIRINOX.

Intervention: Leukapheresis is performed after which monocytes are used for differentiation to dendritic cells. Autologous dendritic cells pulsed with an allogeneic tumor lysate (MesoPher) will be administered intra-dermally and intravenously 3 times every 2 weeks. Booster vaccinations are given after 3 and 6 months. On the same day after administration of MesoPher a CD40 agonist (mitazalimab) will be administered intravenously.

Study parameters/endpoints: The main study endpoint are the dose-limiting toxicities of MesoPher/mitazalimab combination therapy. The secondary endpoints are the induced immune responses on therapy and the radiographical response rate according to RECIST and iRECIST.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Patients have to undergo additional outpatient clinic visits for this study and additional invasive procedures specifically for this trial, e.g. intravenous catheter placement and tumor metastasis biopsies. Although these are invasive procedures, associated risks are limited. Intravenous access is necessary during every visit, i.e. for leukapheresis, for drawing blood samples and for the administration of study medication. Leukapheresis is a standard procedure and will be performed according to our institutional guidelines. Leukapheresis demonstrates a limited risk for transient thrombocytopenia and leukopenia. Previous clinical studies have shown that injection with tumor lysate-pulsed dendritic cells (MesoPher) was well tolerated without major systemic toxicity, with the exception of low-grade flu-like symptoms (REACtiVE Trial, NL67169.000.18; DENIM/MM04: NCT03610360; MM03 NL44330.000.14 / NCT02395679).

Also, intravenous injection of mitazalimab up to 1200 µg/kg was well tolerated with manageable side effects. There are currently no trials investigating this combination therapy. Combining two immunomodulatory drugs increases the risk for toxicity. The objective of this phase I study is to investigate safety and tolerability of administrating MesoPher/mitazalimab combination therapy in metastatic pancreatic cancer patients. Patients may have potential beneficial anti-tumor responses following study medication.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic pancreatic cancer as defined by the presence of radiologically suspect metastatic lesions.
* Inclusion ≤ 4 weeks after stopping FOLFIRINOX chemotherapy.
* No more than 1 line of chemotherapy for metastatic disease is allowed. Prior FOLFIRINOX for locally advanced disease if given within 1 year before screening will be counted as first-line treatment. Any FOLFIRINOX given in the curative intent setting if more than a year before screening will not be considered first line therapy.
* An accessible metastatic lesion for histological tissue collection.
* Patients must be at least 18 years old and must be able to give written informed consent.
* WHO performance status 0-1.
* Patients must have normal organ function and adequate bone marrow reserve: absolute neutrophil count > 1.0 x 109/l, platelet count > 100 x 109/l, and Hb > 6.0 mmol/l (as determined during screening). Transfusion in the 2 weeks preceding screening is not allowed.
* Laboratory tests: ASAT/ALAT <5xULN (upper limit of normal), bilirubine <1.5xULN, Creatinine value <1.5xULN, Lactate dehydrogenase value < ULN and albumin value > LLN (lower limit of normal).
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test just prior to the first study drug administration on Day 1, and must be willing to use an effective contraceptive method (intrauterine devices, hormonal contraceptives, contraceptive pill, implants, transdermal patches, hormonal vaginal devices, infusions with prolonged release) or true abstinence (when this is in line with the preferred and usual lifestyle)* during the study and for at least 12 months after the last study drug administration.

  *True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (such as calendar, ovulation, symptothermal, postovulation methods) and withdrawal are not acceptable methods of contraception.
* Men must be willing to use an effective contraceptive method (e.g. condom, vasectomy) during the study and for at least 12 months after the last study drug administration.
* Ability to return to the hospital for adequate follow-up as required by this protocol.
* Written informed consent according to ICH-GCP.

Exclusion Criteria:

* Medical or psychological impediment to probable compliance with the protocol.
* Abdominal ascites.
* Current or previous use of a CD40 antibody and/or anti-tumor vaccinations.
* Current use of steroids (or other immunosuppressive agents). Patients must have had 6 weeks of discontinuation and must stop any such treatment during the time of the study. Prophylactic usage of dexamethasone during chemotherapy is excluded from this 6 weeks interval.
* Prior malignancy except adequately treated basal cell or squamous cell skin cancer, superficial or in-situ cancer of the bladder or other cancer for which the patient has undergone curative intent treatment and has been disease-free for two years.
* Serious concomitant disease, or active infections.
* History of autoimmune disease, organ allografts or active acute or chronic infection, including but not limited to HIV and viral hepatitis.
* Serious intercurrent chronic or acute illness such as pulmonary disease (asthma or COPD), cardiac disease (NYHA class III or IV), hepatic disease or other illness considered by the study coordinator to constitute an unwarranted high risk for the investigational treatment.
* Known allergy to shell fish (may contain keyhole limpet hemocyanin (KLH)).
* Pregnant or lactating women.
* Inadequate vein access to perform leukapheresis.
* Concomitant participation in another clinical intervention trial (except participation in a biobank study).
* An organic brain syndrome or other significant psychiatric abnormality which would compromise the ability to give informed consent, and preclude participation in the full protocol and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities (DLTs) as assessed by CTCAE v5.0 | From first dose (week 0 of treatment phase) to end of the DLT observation period (week 6 of treatment phase)
  The number of patients experiencing a DLT will be determined. Toxicities will be scored according to CTC criteria version 5.0 (Published November 27th, 2017). The toxicities occurring during 6 weeks after the first vaccination (i.e., the DLT observation period), will be considered as DLT, when considered possibly, probably or definitively related to MesoPher and/or mitazalimab combination therapy. All patients that cannot complete the first 3 doses as planned due to directly related toxicity will be discussed in the Study Steering Committee and they will determine whether the patient is classified as having a DLT.

SECONDARY OUTCOMES:
Determine the presence of vaccine-induced dendritic cell mediated immune responses using ELISA and flow cytometry. | From baseline to end of study (week 36)
  Keyhole Limpet Hemocyanin (KLH) responses: KLH is part of the DC vaccine and is used as a surrogate marker for DC-mediated immune stimulation and persistence of this response. KLH is known to induce a specific adaptive immune response readily detectable in sera (antibody response) and PBMC of vaccinated individuals. Serum samples will be collected before, during and after DC therapy as well as at selected intervals during follow-up. Humoral responses to KLH will be detected using ELISA. In addition, we will also measure cellular responses against KLH. Dendritic cells will be loaded with KLH protein lysate and co-cultured in vitro with PBMCs taken before and after study therapy. After co-culture, T cells will be stained for activation, cytotoxic and degranulation markers and measured by flow cytometry.
Determine the intratumoral treatment effect by measuring T cell influx | From baseline to week 6
  We will use immunohistochemistry to stain T cells in order to determine T cell influx before and after 3 study treatments.
Determine vaccine-induced changes in the frequency of immune cell subsets using flow cytometry | From baseline to end of study (week 36)
  Phenotypical analysis of peripheral blood mononuclear cells (PBMCs) will be conducted with Aurora spectral flow cytometry immune panels comprising 40 different antibodies to analyze changes in the lymphoid and myeloid cell compartments. Vaccine-induced changes in the frequencies of immune cell (subsets) that represent distinct lineages and/or express different levels of activation, differentiation and co-signaling markers are measured. Combination of these readouts allows for the generation of immune profiles for individual patients.
Determining predictive gene expression signatures related to therapy outcome using NanoString technology | From baseline to end of study (week 36)
  Immuno-oncology gene expression signatures will be determined on PBMCs obtained pre- and post-combination treatment and on RNA isolated from OCT-embedded positive DTH skin reactions. This provides us with comprehensive profiling of the immune response including mechanistic pathway activity induced by DC/αCD40 combination therapy.
Radiological response rate as defined by RECIST version 1.1 and iRECIST | From baseline to end of study (week 36)
  Patients undergo regular radiological evaluations until documented evidence of progression as defined by RECIST 1.1 criteria. After each radiographic evaluation patients will be assigned a RECIST response of complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD) depending on the status of their disease compared to baseline and previous assessments. If a patient has had a radiological assessment, which cannot be evaluated, then the patient will be assigned a visit response of not evaluable (NE) (unless there is evidence of progression, in which case the response will be assigned as PD).

CONTACTS AND LOCATIONS:
Overall Officials: Ferry Eskens, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided